CLINICAL TRIAL: NCT04050215
Title: Impact of 68GA-PSMA-11 PET/CT on Initial and Subsequent Treatment Strategies of Patients With Prostate Cancer
Brief Title: 68GA-PSMA-11 PET/CT Scan in Impacting Treatment Strategies for Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-001336; NCI-2019-04439 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Prostate Carcinoma; PSA Level Greater Than Fifty; PSA Progression; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diagnostic (68Ga-PSMA-11 PET/CT) (Experimental): Patients receive 68Ga-PSMA-11 IV and undergo PET/CT scan over 3 hours. Patients may be reenrolled in the study, if 68Ga-PSMA-11 PET/CT is performed for subsequent management decision.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68-labeled PSMA-11; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the impact of 68GA-PSMA-11 positron emission tomography (PET)/computed tomography (CT) scan on treatment strategies for patients with prostate cancer. Diagnostic imaging procedures, such as 68GA-PSMA-11 PET/CT scan, may help doctors plan the best treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the impact of gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) PET/CT on initial and subsequent treatment strategies of patients with prostate cancer.

OUTLINE:

Patients receive 68Ga-PSMA-11 intravenously (IV) and undergo PET/CT scan over 3 hours. Patients may be reenrolled in the study, if 68Ga-PSMA-11 PET/CT is performed for subsequent management decision.

After completion of study, patients are followed up within 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill criteria for initial staging or restaging as outlined below:

  * Initial treatment strategy decisions (initial staging): All patients with histologically proven prostate cancer or strong suspicion of prostate adenocarcinoma based on very high prostate-specific antigen (PSA) levels (> 50 ng/mL) who require an initial treatment/management decision who may be candidate for any of the following strategies:

    * Surgery
    * External radiation therapy (RT)
    * Other focal therapies
    * Systemic medical treatment
    * Watchful waiting
  * Assessment for subsequent treatment strategy (restaging), any of the following:

    * Patients with biochemical recurrence who are potential candidates for any salvage treatment. Biochemical recurrence is defined by rising PSA after definitive therapy with prostatectomy or radiation therapy, as any of the following:

      * Post radical prostatectomy (RP): PSA equals to or greater than 0.2 ng/mL measured more than 6 weeks after RP
      * Post-radiation therapy: Nadir + greater than or equal to 2 ng/mL rise in PSA
    * Patients with known prostate cancer who undergo restaging because of new symptoms
    * Patients with known metastatic prostate cancer who undergo restaging because of rising PSA with negative or inconclusive conventional imaging
    * Patients with known prostate cancer who are treated medically or with radioligand therapy (RLT) in whom response to treatment is assessed
    * Note: Patients may be reenrolled in the study, if 68Ga-PSMA PET/CT is performed for subsequent management decision
* Capability to provide written informed consent
* Able to remain still for duration of each imaging procedure (about 30 minutes)

Exclusion Criteria:

* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance
* Inability to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 937 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Intended and implemented management changes after gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) positron emission tomography (PET)/computed tomography (CT) | Up to 3-6 months after completion of imaging
  A separate analysis of initial versus subsequent management will be performed. Will be evaluated using descriptive statistics for both the treatment modality analysis and the disease stage based management analysis. Questionnaires will be collected to determine the intended patient management before and intended management changes after PET/CT, and to determine whether intended management changes were implemented. The outcome measure is the rate of change (%) as assessed by the questionnaires before and after PET.

SECONDARY OUTCOMES:
Prognostic value of the 68Ga-PSMA-11 PET/CT miTNM classification for biochemical progression-free survival (PFS) | From inclusion to date until PSA progression or death (whichever occurs first), assessed up to 12 months
Prognostic value of the 68Ga-PSMA-11 PET/CT miTNM classification for radiographic PFS | From inclusion to date until first site of disease is found to progress or death (whichever occurs first), assessed up to 12 months
  Nodal and visceral disease will be evaluated on cross-sectional imaging using Response Evaluation Criteria in Solid Tumors 1.1/Prostate Cancer Working Group 3 (PCWG3) criteria. Bone metastases will be evaluated using bone scintigraphy and new lesions have to be confirmed on a second scan (2+2 rule) using PCWG3 criteria.
Prognostic value of the 68Ga-PSMA-11 PET/CT miTNM classification for overall survival | From inclusion to date of death, assessed up to 12 months
Positive predictive value (PPV) on a per-patient and per-region basis of 68Ga-PSMA-11 PET for detection of tumor location | Up to 12 months
  Confirmed by histopathology/biopsy or follow-up assessed separately for initial staging and restaging. Will be calculated and reported along with the corresponding two-sided 95% confidence intervals. The confidence intervals will be constructed using the Wilson score method. PPV will be reported for each of the three blinded readers independently. Detection rates on a per-patient basis of 68Ga-PSMA-11 PET stratified by prostate-specific antigen (PSA) value will be summarized in tabular format and compared between PSA strata using chi-square analysis. Detection rate is defined as number of patients with PSMA positive disease, independent of pathology, imaging or clinical follow-up. A detection rate will be reported for each reader independently stratified by PSA.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Ma TM, Gafita A, Shabsovich D, Juarez J, Grogan TR, Thin P, Armstrong W, Sonni I, Nguyen K, Lok V, Reiter RE, Rettig MB, Steinberg ML, Kupelian PA, Yang DD, Muralidhar V, Chu C, Feng F, Savjani R, Deng J, Parikh NR, Nickols NG, Elashoff D, Czernin J, Calais J, Kishan AU. Identifying the Best Candidates for Prostate-specific Membrane Antigen Positron Emission Tomography/Computed Tomography as the Primary Staging Approach Among Men with High-risk Prostate Cancer and Negative Conventional Imaging. Eur Urol Oncol. 2022 Feb;5(1):100-103. doi: 10.1016/j.euo.2021.01.006. Epub 2021 Feb 16. PMID 33602654